CLINICAL TRIAL: NCT01659775
Title: A Multicenter, Randomized, Open-label, Paralleled-group, Active-controlled, Phase IV Study to Evaluate the Efficacy and Safety of Sancuso Patch (Granisetron) in Chemotherapy-induced Nausea and Vomiting (CINV) Associated With the Administration of Highly Emetogenic (HE) Chemotherapy
Brief Title: Phase 4 Trial to Evaluate the Efficacy and Safety of Sancuso Patch in Chemotherapy-induced Nausea and Vomiting Associated With the Administration of Highly Emetogenic Chemotherapy (HEC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-SCSCL001
Record Dates: First submitted 2012-07-27; First posted 2012-08-08 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2012-01

CONDITIONS: Chemotherapy-induced Acute or Delayed Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sancuso patch (Experimental)
  Interventions: Drug: Sancuso patch
- Zofran (Active Comparator)
  Interventions: Drug: Zofran inj.+Zofran tab.

INTERVENTIONS:
Drug: Sancuso patch — Eligible patients were randomized to Sancuso patch or Zofran groups and received the assigned treatment for 5days.
  Experimental arm: Sancuso patch (34.3mg) applied to upper, outer arm 2days (48-24hours) prior to start of chemotherapy.
  Arms: Sancuso patch
Drug: Zofran inj.+Zofran tab. — Eligible patients were randomized to Sancuso patch or Zofran groups and received the assigned treatment for 5days.
  Active Comparator arm: administered intravenously (24mg or 32mg) on Day 1 of chemotherapy and orally (8mg bid) on Day 2-5.
  Arms: Zofran

SUMMARY:
This is a multicenter, randomized, open-label, paralleled-group, active-controlled study.

The study is to demonstrate non-inferiority of the Granisetron Transdermal Delivery System (GTDS) efficacy compared with the ondansetron efficacy with regard to Complete Response (CR) of Chemotherapy Induced Nausea and Vomiting (CINV).

Patients scheduled to receive the one cycle of a HE chemotherapy regimen administered for 1-5 days will attend a Screening Visit 2 to 14 days before start of HE chemotherapy. Eligible patients will be randomized to 1 of 2 treatment groups at the Randomization Visit (1 to 2 days prior to HE chemotherapy).

* Sancuso patch
* Zofran inj. + Zofran tab.

The patch will be applied 2days (48-24h) prior to first daily dose of the highly emetogenic chemotherapy regimen and remain in place for 5 days after start of chemotherapy. The patient will be assessed daily until 5days after first chemotherapy administration. Adverse Events (AEs) will be collected until 2 days after the final dose of IP. Non-serious AEs will be followed-up until 2 days after the final dose of IP. Serious adverse events will be followed-up until they are resolved, stable or until the patient is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 20 yrs
2. Eastern Cooperative Oncology Group performance status 0, 1, 2
3. Life expectancy of ≥ 3 months
4. Assigned to receive a cycle of high emetic (HE) chemotherapy regimen including the daily administration of a cytotoxic regimen with the emetogenic potential of level 5 (Hesketh Classification)
5. Patients who signed the informed consent form

Exclusion Criteria:

A. Previous History

1. Hypersensitivity to adhesive plasters
2. Contraindications to 5-HT3 receptor antagonists
3. Any other relevant medical history (at the discretion of the investigator)

B. Concomitant Medical Condition

1. Current alcohol, drug or medication abuse
2. Currently pregnant or breast feeding women, including planning pregnancy
3. Clinically relevant abnormal laboratory values (at the discretion of the investigator)
4. Clinically relevant hepatic, renal, infectious, neurological or psychiatric disorders, or any other major systemic illness (at the discretion of the investigator)
5. Any cause for nausea and vomiting other than CINV
6. Any episode of retching, vomiting or uncontrolled nausea in the 72 h period prior to the chemotherapy administration
7. Clinically relevant abnormal ECG parameters at the discretion of the investigator

C. Concomitant Therapy/Medication

1. Concomitant radiotherapy of total body, brain or upper abdomen within one week of study entry or planned during the study
2. Intake of medication to control the symptoms of a brain tumour, brain metastasis or seizure disorder or neuropathy (unless peripheral neuropathy at the discretion of the investigator)
3. Patients using selective serotonin reuptake inhibitor (SSRI) antidepressants (unless a stable dose for the duration of the study)
4. Receipt of a narcotic analgesics (acceptable at the discretion of the investigator)
5. Receipt of any other investigational drug < 30 days before the study start or during the study
6. Scheduled to receive a neurokinin NK1 receptor antagonist, dopamine receptor antagonist or another 5-HT3 receptor antagonist at 72 h prior to the administration of the chemotherapy or scheduled to do those medication after patch removal
7. Drugs known to increase the QTc interval (unless a stable dose for the duration of the study at the discretion of the investigator)

D. Other

1. Patients unlikely to comply with the study protocol (at the discretion of the investigator), e.g. uncooperative attitude, inability to return for follow-up visits and unlikelihood of completing the study
2. The patch adhesion level was not more than 50% on the day of chemotherapy or the patch was not attached within two days before the chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The percentage of patients achieving Compete Response (CR) without rescue therapy from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen

SECONDARY OUTCOMES:
The percentage of patients achieving Complete Response (CR) | overall (Day 1~5)
The percentage of patients achieving Complete Control (CC) without rescue therapy from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen
The percentage of patients achieving Compete Control (CC) | overall (Day 1~5)
severity of nausea | overall (Day 1~5)
severity of vomiting | overall (Day 1~5)
Frequency of nausea from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen
Frequency of vomiting from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the chemotherapy regimen
Patient's satisfaction with anti-emetic therapy | overall (Day 1~5)
  The overall response to anti-emetic therapy was assessed and recorded by patients at Visit 8. The patient was asked to evaluate his/her satisfaction with the control of nausea and vomiting by marking the FLI-E (Functional Living Index - Emesis) with vertical lines.
The percentage of patients achieving Complete Response (CR) | per day (Day1, 2, 3, 4, 5)
The percentage of patients achieving Compete Control (CC) | per day (Day 1, 2, 3, 4, 5)
severity of nausea | per day (Day 1, 2, 3, 4, 5)
severity of vomiting | per day (Day 1, 2, 3, 4, 5)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hyoung Kang, MD,PhD, Principal Investigator — Seoul St'. Mary's Hospital; Hoon-Kyo Kim, MD,PhD, Principal Investigator — St Vincent's Hospital; Suk-Young Park, MD,PhD, Principal Investigator — Daejeon St. Mary's hospital; Jong-Youl Jin, MD,PhD, Principal Investigator — Bucheon St. Mary's Hospital; In-Sook Woo, MD,PhD, Principal Investigator — Yeouido St. Mary's Hospital; Yoon-Ho Ko, MD,PhD, Principal Investigator — Uijeongbu St. Mary's Hospital; Der-Sheng Sun, MD,PhD, Principal Investigator — Cheongju St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea